CLINICAL TRIAL: NCT02479659
Title: A Cluster Randomised Trial on the Impact of Integrating Early Infant HIV Diagnosis With the Expanded Programme on Immunization on Immunization and HIV Testing Rates in Rural Zambian Health Facilities
Brief Title: Measuring the Impact of Integrating Maternal and Newborn HIV Testing With Childhood Immunization Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IDinsight (Other)
Collaborators: Zambia Center for Applied Health Research and Development (Other); Ministry of Health, Zambia (Other Government); Minister of Community Development, Mother and Child Health, Zambia (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2015-06-14; First posted 2015-06-24 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: HIV
Keywords: Immunizations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Facilities in this arm maintained status quo HIV testing and routine childhood immunization services
- Simple Intervention (Experimental): This included: 1) HIV testing commodity reinforcement and 2) a policy reinforcement meeting
  Interventions: Other: HIV testing commodity reinforcement; Other: Policy reinforcement meeting
- Comprehensive Intervention (Experimental): This arm included: 1) HIV testing commodity reinforcement, 2) a policy reinforcement meeting, 3) community sensitization, 4) Opt-out HIV testing for mothers and newborns, and 5) Operational support for service integration
  Interventions: Other: HIV testing commodity reinforcement; Other: Policy reinforcement meeting; Other: Opt-out HIV testing for mothers and newborns; Other: Operational support for service integration; Other: Community sensitization

INTERVENTIONS:
Other: HIV testing commodity reinforcement — HIV testing commodities were replenished directly (outside of the government supply) in the event of a stock-out by study staff. Treatment facilities were visited monthly to assess stock levels, and facility staff could contact study staff when stock levels were low.
  Arms: Comprehensive Intervention; Simple Intervention
Other: Policy reinforcement meeting — District health officials met with facility staff to remind them of the current HIV testing policies for mothers and newborns in Zambia. Current policy states mothers with unknown or previously negative status should be tested every 3 months until the infant is 18 months of age. HIV-exposed newborns should be tested at 6 weeks and 6 months.
  Arms: Comprehensive Intervention; Simple Intervention
Other: Opt-out HIV testing for mothers and newborns — Facility staff were instructed to examine the maternal HIV status on the under-five (U-5) or antenatal care (ANC) card for all infants attending their first U-5 visit and do the following:
  * If marked Confirmed Exposed (CE), the health care worker conducted the DBS test on the infant only.
  * If marked, Mother Status Unknown (MSU) or Confirmed Not Exposed (CNE) the mother or caregiver was asked if the mother had ever tested HIV-positive. If yes, a DBS was done on the infant only. If no, the mother was offered an HIV antibody test in an opt-out manner.
  Arms: Comprehensive Intervention
Other: Operational support for service integration — The evaluation team worked with facility staff to identify efficient allocations of staff and tailor the order of services. A key component of the operational optimization was a new patient triaging approach that sorted patient U-5 cards into bins and used separate queues for three types of patients: 1) first visit infants (six weeks), 2) second visit or later infants who required immunizations and 3) infants who were scheduled to only receive growth monitoring.
  Arms: Comprehensive Intervention
Other: Community sensitization — Health facility staff were instructed to communicate all aspects of the Comprehensive Intervention during ANC appointments, in-facility child birth deliveries, and postnatal care (PNC) visits. Additionally, at six week immunization visits, mothers and caregivers received group counseling on opt-out HIV screening service and the importance of regular HIV screening for mother and child health. Finally, the research team engaged Safe Motherhood Action Groups (SMAGs), community health workers (CHWs), and active neighborhood health committee members to further increase awareness in facility catchment areas. These community members completed low-touch community sensitization over changes that would be made to U-5 services.
  Arms: Comprehensive Intervention

SUMMARY:
This randomized evaluation measured the impact of two levels of support for the integration of infant and postpartum maternal HIV testing with routine immunization services in Southern Zambia on the number of postpartum maternal HIV tests, infant HIV tests, and 1st dose diphtheria, pertussis, and tetanus (DPT1) vaccines.

DETAILED DESCRIPTION:
This evaluation assessed two levels of support for the integration of early infant and maternal HIV testing with existing routine immunization services in rural health facilities in Southern Zambia with the aim of determining whether infant and postpartum maternal HIV testing rates would increase without harming immunization uptake. The evaluation randomized 60 health facilities to one of three study arms: 1) Control (status quo); 2) Simple Intervention; and 3) Comprehensive Intervention. The Simple Intervention included restocking of HIV test kits and reminding health facilities of existing HIV testing guidelines by government health officials. The Comprehensive Intervention included the Simple Intervention components, as well as community sensitization, hands-on operational support to integrate services and improve patient flow, and opt-out HIV testing for mothers and infants according to existing guidelines. The change in the average number of monthly HIV tests and immunizations (DPT1) between the intervention period and baseline were compared between treatment and control facilities.

ELIGIBILITY:
Note that this evaluation used administrative data - no participants were enrolled for the main part of this study. Participants were enrolled for the qualitative portions of the study.

Inclusion Criteria:

* Mothers who had an infant within the past 18 months during the intervention period (Oct 2013 - Mar 2014)
* Infants who were at least six weeks of age and under six months of age during the intervention period (Oct 2013 - Mar 2014)
* Qualitative activities included facility staff and mothers and caregivers whose infants were due for their 6 week immunization during the intervention period.

Exclusion Criteria:

* Mothers who did not have an infant within the past 18 months during the intervention period
* Infants who were less than six weeks of age during the intervention period or greater than six months of age throughout out the intervention period.
* Adults who were not mothers or caregivers with an infant due for his/her 6 week immunization during the intervention period were excluded from the qualitative activities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in average monthly number of infant DBS HIV tests | Baseline and 6 mos (endline)
  Using a difference-in-differences analytic approach, the investigators analyzed counts of the number of infant dried blood spot (DBS) HIV tests administered per month at each of the 60 study facilities between Oct 2013 and Mar 2014 (intervention period), and compared it to retrospective baseline data from Jan 2012 - Sept 2013
Change in average monthly number of maternal postpartum HIV tests | Baseline and 6 mos (endline)
  Using a difference-in-differences analytic approach, the investigators analyzed counts of the number of maternal postpartum HIV tests administered per month at each of the 60 study facilities between Oct 2013 and Mar 2014 (intervention period), and compared it to retrospective baseline data from Jan 2013 - Sept 2013
Change in average monthly number of DPT1 doses administered | Baseline and 6 mos (endline)
  Using a difference-in-differences analytic approach, the investigators analyzed counts of the number of first dose diphtheria, pertussis, and tetanus vaccine (DPT1) administered per month at each of the 60 study facilities between Oct 2013 and Mar 2014 (intervention period), and compared it to retrospective baseline data from Jan 2012 - Sept 2013

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wang, MPAID/MBA, Principal Investigator — IDinsight

REFERENCES:
- [Derived] Wang PC, Mwango A, Moberley S, Brockman BJ, Connor AL, Kalesha-Masumbu P, Mutembo S, Bweupe M, Chanda-Kapata P, Biemba G, Hamer DH, Chibuye B, McCarthy E. A Cluster Randomised Trial on the Impact of Integrating Early Infant HIV Diagnosis with the Expanded Programme on Immunization on Immunization and HIV Testing Rates in Rural Health Facilities in Southern Zambia. PLoS One. 2015 Oct 29;10(10):e0141455. doi: 10.1371/journal.pone.0141455. eCollection 2015. PMID 26513240